CLINICAL TRIAL: NCT05743920
Title: Efficacy of Self-help Forest Bathing (Shinrin-yoku) on Depression, Anxiety, and Stress: A Pilot Randomized Controlled Trial
Brief Title: Self-help Forest Bathing (Shinrin-yoku) on Depression, Anxiety, and Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PSY030
Record Dates: First submitted 2023-02-16; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Depression, Anxiety; Stress
Keywords: Lifestyle medicine; Randomised controlled trial; Depression; Stress; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-help Forest Bathing Group (Experimental): Participants in the FB group will perform forest bathing activity at the Chinese University of Hong Kong for two session.
  Interventions: Behavioral: Self-help Forest Bathing
- Wait List Group (Other)
  Interventions: Behavioral: Self-help Forest Bathing

INTERVENTIONS:
Behavioral: Self-help Forest Bathing — The self-help forest bathing includes two sessions (i.e., participants will perform the first intervention within week 1 to 3, and the second intervention within week 4 to 6) that are related to the following forest bathing activities : (a) forest meditation, (b) forest walking, (c) calling attention to sensory experiences of the forest, including seeing, hearing, touching, and smelling, and (d) building connection to the nature by partnership invitation. Each session will last for 45 minutes.

SUMMARY:
The objective of this pilot randomized controlled trial is to evaluate the efficacy and acceptability of self-help forest bathing on depression, anxiety, and stress in the Hong Kong adult population.

Prior to all study procedures, eligible participants will be required to complete an online informed consent form (with telephone support). Around 80 eligible participants aged between 18 to 65 years old with at least a mild level of depression, anxiety, or stress symptoms will be randomly assigned to either the self-help forest bathing intervention group (FB group) or the waitlist control group (WL group) in a ratio of 1:1.

Participants in the FB group will receive forest bathing guidance via an in-house smartphone app. The WL group will be asked to maintain their typical activity in week 1-7. This group will receive the guide upon trial completion in week 8.

The outcomes of the interest will include generalized anxiety symptoms, depressive symptoms, insomnia symptoms, wellbeing, health-related quality of life, functional impairment at baseline (week 0), immediate (week 7), and 1-month post-intervention assessments (week 10). Treatment credibility and acceptability will be collected at baseline and immediately after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents;
2. Aged between 18 to 65 years;
3. Meet the threshold for mild depression (score of >5 on the Patient Health Questionnaire 9 [PHQ-9], anxiety (>5 Generalized Anxiety Disorder 7 [GAD-7]), or stress (>15 on the Depression, Anxiety, and Stress Scale [DASS-21] stress subscale, after multiplying score by 2);
4. Able to read and understand Chinese and type in Chinese or English
5. Have an Internet-enabled mobile device (iOS or Android operating system)
6. Willing to provide informed consent and comply with the trial protocol

Exclusion Criteria:

1. Received psychotherapy for depression, anxiety and stress in the past 6 months;
2. A change in psychotropic drugs or over-the-counter medications that target depression, anxiety, and stress within 2 weeks before the baseline assessment.
3. Patient Health Questionnaire-9 (PHQ-9) item 9 score > 2, indicating a moderate level of suicidal risk that requires active crisis management (referral information to professional mental health services will be provided);
4. Currently participating in another intervention study that may potentially affect mental health;
5. Self-disclosure of having unsafe health conditions for which physical activity was contraindicated by physicians;
6. Self-disclosure of any psychiatric, medical, or neurocognitive disorder(s) that makes participation unfeasible;
7. Pregnancy;
8. Hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, immediate post-treatment, and 1-month follow-up
  The PHQ-9, a 9-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Baseline, immediate post-treatment, and 1-month follow-up
  The GAD-7, a 7-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of anxiety over the past two weeks on a 4-point scale, "0" (not at all) to "4" (nearly every day).
Change in the Perceived Stress Scale (PSS) | Baseline, immediate post-treatment, and 1-month follow-up
  The PSS, a 10-item questionnaire measuring the perceived degree of stress across situations over the past month. Items include how unpredictable, uncontrollable, and overloaded do the respondents perceive. The score ranges from "0" (never) to "4" (very often).
Change in the Insomnia Severity Index (ISI) | Baseline, immediate post-treatment, and 1-month follow-up
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the The World Health Organisation- Five Well-Being Index (WHO-5) | Baseline, immediate post-treatment, and 1-month follow-up
  WHO-5 is a short and generic global rating scale measuring subjective well-being.
Change in the Sheehan Disability Scale (SDS) | Baseline, immediate post-treatment, and 1-month follow-up
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline and immediate post-treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success. Specific wording referencing "anxiety" was changed to refer to "depression".
Change in the Treatment Acceptability and Adherence Scale (TAAS) | Baseline and immediate post-treatment
  TAAS is a self-reported, ten-item questionnaire that is rated by a seven-point Likert scale from 1 to 7, and it aims at evaluating the clients' attitude toward the treatment sessions by four domains, including acceptability, adherence, drop-out, and distress. Specific wording referencing "anxiety" was changed to refer to "depression".
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediate post-treatment, and 1-month follow-up
  A preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The SF-6D index, scored from 0.0 (worst health state) to 1.0 (best health state)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Yan-Yee Ho, Study Chair — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No